CLINICAL TRIAL: NCT06098040
Title: Long-Term Feedback Effect of Flash Glucose Monitoring (Freestyle Libre2®) in Newly-Diagnosed Type 2 Diabetic Patients: a Randomized Monocentric Parallel-group Clinical Trial
Brief Title: Long-Term Feedback Effect of FGM in Newly-Diagnosed T2D Patients
Acronym: DIAFLASH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Silvia Manfrini, Principal Investigator and head of the endocrinology and diabetes unit, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIAFLASH
Record Dates: First submitted 2023-10-04; First posted 2023-10-24 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
Keywords: time in range; quality of life; bio feedback; flash glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: three-armed parallel group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- group 2 - FGM continuous (Experimental): Patients will be asked to wear the sensor FreeStyle Libre2 continuously
  Interventions: Device: flash glucose monitoring continuous
- group 3 - FGM intermittent (Experimental): will be asked to wear the sensor FreeStyle Libre2 intermittently
  Interventions: Device: flash glucose monitoring intermittent
- group 1- SMBG (Active Comparator): Patients will be asked to test capillary blood glucose as recommended by subjects' usual provider
  Interventions: Diagnostic Test: capillary blood test

INTERVENTIONS:
Device: flash glucose monitoring continuous — Group 2 (FGM continuous): will be asked to wear the sensor FreeStyle Libre2 for the FGM with the following frequency fashion continuously for the first 12 weeks and followed by 12 weeks testing as recommended by their usual provider.
  Arms: group 2 - FGM continuous
Diagnostic Test: capillary blood test — Group 1 (SMBG): will be asked to test capillary blood glucose as recommended by subjects' usual provider for the first 12 weeks and followed by 12 weeks testing as recommended by their usual provider.
  Arms: group 1- SMBG
Device: flash glucose monitoring intermittent — Group 3 (FGM intermittent): will be asked to wear the sensor FreeStyle Libre2 for the FGM with the following frequency fashion 1 week off/2 weeks on for the first 12 weeks and followed by 12 weeks testing as recommended by their usual provider.
  Arms: group 3 - FGM intermittent

SUMMARY:
This clinical trial aims to evaluate the educational training of 12-weeks using flash glucose monitoring (FGM) FreeStyle Libre2 (FSL2; Abbott Diabetes Care Inc., Alameda, CA, USA) in newly- diagnosed T2D subjects who are treated with metformin in term of sustained improvement in glycemic variability (TIR) after the discontinuation of FGM compared to self-monitoring of blood glucose (SMBG). This clinical trial also aim to explore which frequency of sensor wear at the diagnosis is more effective in achieving a sustained improvement in TIR after the FGM discontinuation over time.

DETAILED DESCRIPTION:
Diabetes self-management represents the cornerstone of successful and cost-effective diabetes care, reducing the occurrence of complications, hospital admissions and readmission as well as estimated lifetime health care costs related to a lower risk for complications. Recent advances in diabetic technology may help to address some of these issues : Flash glucose monitoring (FGM) is a novel system of interstitial glucose monitoring intended to replace the capillary blood glucose measurement which proved to ameliorate glycemic variability and quality of life, beyond the good precision, increased time in range, and ease of wear. However, FGM is not currently used as an educational tool in patients with newly diagnosis of T2D who are not on insulin therapy.

Therefore, the rationale for this three-armed parallel group randomized controlled trial is that the continuous flow of data from FGM and the visual display of moment-to-moment glucose levels as a trend could provide real-time feedback also in newly T2D patients, assessing which frequency of sensor is superior in enhancing mindfulness and in ameliorating of glycemic control ,quality of life and well-being perception.

The entire study participation will span approximately 6 months and will be performed in the facilities of Fondazione Policlinico Campus Bio-Medico University of Rome enrolling 42 participants. The intervention phase will last 12 weeks followed by more 12 weeks in the follow-up phase. Each participant will have a screening visit ( week -4), a baseline visit ( week -2), a randomization visit (week 0) and three follow up visits at week 12 and 23 and 24 for all the groups.

Every group will wear also a blinded device (Free Style Libre Pro IQ) for registration of glicemyc variability at the baseline visit and a the end of the study ; group 1 will wear it also between intervention and follow-up phase ( weeks 11-12).

All patients will be asked to fill out a food diary at both the intervention and follow-up phases. A high glycemic index meal will also be administered during the randomization visit ( week 0) in order to record the emotional state of study subjects in response to postprandial glycemic values. Randomization will be performed following a ratio equal to 1:1:1 and blocked for gender.

The primary outcome of the study is the difference in the means of time in range (TIR) at weeks 23-24 adjusted for baseline phase values. Secondary endpoints include the difference in TIR assessed at weeks 11-12 among the three groups and within the three groups as well as difference in A1c, HOMA IR, weight, body composition and oxidative stress among the groups. Quality of life/well-being perception/mindfulness will be investigated at week 0, week 12 and week 24 through several questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus ( according to the ADA Guidelines ) within the past 12 months
* Must be taking only metformin as glucose lowering treatments,
* Older than 18 years,
* Body Mass Index equal or greater than 25 Kg/m^2,
* Must be able to provide written informed consent .

Exclusion Criteria:

* diagnosis of type 1 diabetes;
* glycated hemoglobin exceeding 8.5%
* alcohol or drug abuse/dependency
* antidiabetic therapy other than metformin;
* pregnancy (on-going or planned during the study);
* severe illness (physical or mental health);
* cognitive impairment;
* high dose steroids;
* hospitalized more than 2 times in past 12 months
* previous bariatric intervention or gastrectomy;
* pace maker use
* uncorrected vision impairment;
* already using a continuous glucose monitor or flash glucose monitor;
* any allergy to the component of the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 1:1
Enrollment: 42 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
time in range | 6 months
  difference in the means of time in range (TIR) registered at the weeks 23-24 phase through blinded device Free style Libre PRO-IQ, among the three groups and adjusted for baseline phase values.

SECONDARY OUTCOMES:
time in range | 3 months
  difference in the means of time in range (TIR) assessed at weeks 11-12 among the three groups,and adjusted for baseline phase values
mindfulness | 3-6 months
  changes in eating mindfulness questionnaire score ( 28 items, each questions from 0 to 4 points) evaluated among the three groups and adjusted for baseline values. Higher scores on the mindful eating questionnaire overal, and on each of the categories ( Awareness , Distraction,Disinhibition,Emotional Response, External Cues)-has been associated with a lower body mass index and long-term weight maintenance
Body Mass Index (BMI,kg/m^2) | 6 months
  changes in body mass (Kg) divided by the square of the body height (m), and is expressed in units of kg/m^2, resulting from mass in kilograms (kg) and height in metres (m) at weeks 12 and 24.
Body Composition | 6 months
  changes in fat mass ( Kg ) and Fat free mass (Kg) assessed with bioelectrical Impedance Analysis adjusted for baseline values.
Physical activity | 6 months
  evaluation of the types of intensity of physical activity in the previous 7 days assessed by th International Physical Activity Questionnaire ( IPAQ)- short form at week 24 among the three groups. Total physical activity will be expressed in MET ( Metabolic Equivalent of Task)-min/week and time spent sitting . MET< 700 is indicative of inactive person, MET above 2520 is indicative of very active person
d-ROMs derivatives-reactive oxygen metabolites | 3-6 months
  changes in derivatives-reactive oxygen metabolites (d-ROMs, U.Carr) after the discontinuation of FGM compared with SMBG
PAT plasma antioxidant capacity | 3-6 months
  changes in plasma antioxidant capacity ( PAT test, μmol/L ) after the discontinuation of FGM compared with SMBG

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Manfrini, MD, Principal Investigator — Campus Bio-Medico University; Rossella Tozzi, MD PhD, Study Chair — Campus Bio-Medico University; Dario Tuccinardi, MD PhD, Study Director — Campus Bio-Medico University
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication on request
Supporting Information: Study Protocol, CSR
Time Frame: after the publication
Access Criteria: IPD that underlie results in a publication on request